CLINICAL TRIAL: NCT02629016
Title: Stress Reduction: A Pilot Study With Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Jeanette Johnstone, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00011301
Record Dates: First submitted 2015-12-08; First posted 2015-12-11 (Estimated); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Physiological Stress; Psychological Stress
MeSH Terms: conditions — Stress, Psychological | interventions — Mindfulness; Health

ARMS (3):
- Mindfulness (Experimental): Education and experiential exercises for mindfulness including movement, thoughts and meditation
  Interventions: Other: Mindfulness
- Wellness (Active Comparator): Education and experiential exercises for general wellness including sleep hygiene, goal setting and power poses.
  Interventions: Other: Wellness
- Waitlist (No Intervention): Students receive regular health class instruction without intervention.

INTERVENTIONS:
Other: Mindfulness
  Arms: Mindfulness
Other: Wellness
  Arms: Wellness

SUMMARY:
This study will evaluate the feasibility of providing an onsite mindfulness intervention, delivered as part of the school health curriculum, to help high school-attending adolescents cope with stress.

DETAILED DESCRIPTION:
For this study, sophomores who are enrolled in health at Jesuit High School, (n = 320 students) will be invited to participate in a research study, conducted during health class, comparing mindfulness to a wellness or waitlist control. The students will be randomized by classroom, to either wellness or mindfulness or waitlist, with approximately 3-4 classes per intervention or control. Initially, six classes or sections of health will be randomized to one of the two active interventions, with the remaining classes/sections of health on the waitlist. Both of the intervention groups will meet weekly, during one of the regularly scheduled health classes, and have daily assignments. The students in the waitlisted classrooms will receive an intervention at the start of the next term. At the end of the study, students will have access to the materials from the other group, if desired.

ELIGIBILITY:
Gender:

•Both: both female and male participants are being studied

Age for students:

•Minimum age 13 year, 0 months; •Maximum:16 years, 0 months

Age for parents:

N/A°

Inclusion Criteria:

Adolescents who are enrolled in health class at Jesuit High School,

* Who have access to an iPad, cell phone or computer,
* Are considered reliable and compliant with the study protocol including willing to abide by randomization process, willingness to commit to daily practice activities for the duration of the study.
* Students taking psychiatric medication including stimulants, anti-depressants or anxiolytics are eligible to participate provided they are stable on their current dose of medication, have been taking it for at least two weeks, and will remain on the same dose for the remainder of the study. Any changes in medication will be noted.

Exclusion:

* Intellectual disability, as reported by parent or teacher;
* Current manic episode
* Psychotic episode
* Untreated Post Traumatic Stress Disorder, identified through parent or student report.

Exclusion Criteria:

-

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2015-09; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Depression Anxiety and Stress Scale (DASS) | Change in DASS score from baseline (week 0) to post-intervention (week 9)
  Baseline to post-intervention or waitlist DASS change score
Conners 3 Short Form | Change score from baseline (week 0) to post-intervention (week 9) on Conners
  Baseline to post-intervention or waitlist Conners change score
Automatic Thoughts Questionnaires (ATQ) | Change score from baseline (week 0) to post-intervention (week 9) on ATQ
  Baseline to post-intervention or waitlist ATQ change score

SECONDARY OUTCOMES:
Sleep Quality | Change score from baseline (week 0) to post-intervention (week 9) on sleep
  Baseline to post-intervention or waitlist sleep change score
Stress Reactivity | Change score from baseline (week 0) to post-intervention (week 9) in beats per minute
  Change score from baseline to post intervention or waitlist on heart rate/pulse
Five Factor Mindfulness Questionnaire (FFMQ) | Change score from baseline (week 0), post-intervention (week 9) on FFMQ
  Change in FFMQ score from baseline to post-intervention or waitlist
Stress reactivity | Change score from baseline (week 0) to post-intervention (week 9) blood pressure (BP) sys/dia measurement
  Change score from baseline to post intervention or waitlist on BP
Self-report stress on behavioral tasks | Change score from baseline (week 0) to post-intervention (week 9) on self-rated stress (0-10 likert scale)
  Change from baseline to post-intervention or waitlist on self-reported stress following behavioral tasks
Perceived Stress Scale (PSS) | Change score from baseline (week 0) to post-intervention (week 9) on PSS
  Baseline to post-intervention or waitlist PSS change score

CONTACTS AND LOCATIONS:
Overall Officials: Joel Nigg, PhD, Principal Investigator — OHSU, Psychiatry